CLINICAL TRIAL: NCT06968390
Title: Perinatal Accelerated iTBS Neuromodulation Therapy
Brief Title: Accelerated TMS for Perinatal Depression
Acronym: PAiNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joseph J. Taylor, MD, PhD, Clinical Director of TMS, Center for Brain Circuit Therapeutics, Assistant Professor of Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025P001058; Women's Brain Initiative (Other Grant/Funding Number: Brigham and Women's Hospital)
Record Dates: First submitted 2025-05-02; First posted 2025-05-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-05

CONDITIONS: Perinatal Depression; Post Partum Depression; Major Depressive Disorder
Keywords: TMS; Accelerated TMS; Perinatal Depression; Perinatal; Postpartum; Postpartum Depression; Major Depressive Disorder; Pregnant
MeSH Terms: conditions — Depression, Postpartum; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Open-label aiTBS for pregnant/postpartum individuals (Experimental): 10 iTBS treatment sessions per day (18,000 pulses/day) for 5 consecutive days (90,000 pulses total) to the dorsolateral prefrontal cortex (DLPFC). In the unlikely event that a participant is late for an hourly treatment, then the treatment will be delayed accordingly. The minimum gap between treatments will be 25 minutes. Each iTBS treatment will consist of 60 cycles of 10 bursts of three pulses at 50 Hz delivered in 2-second trains (5 Hz) with an 8-second intertrain interval. Stimulation will be delivered at 90% resting motor threshold (rMT), adjusted for depth of the identified functional connectivity target or based on traditional scalp measurements.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Non-invasive form of brain stimulation.
  Other Names: TMS; Accelerated intermittent theta burst stimulation; aiTBS

SUMMARY:
We are studying a treatment for depression called accelerated Transcranial Magnetic Stimulation (TMS) among pregnant and postpartum individuals. TMS is a focal, non-invasive form of brain stimulation that is cleared by the Food and Drug Administration for depression. Typically, traditional TMS involves daily treatments for 6-8 weeks. In this study, we will offer an accelerated form of TMS that involves multiple daily treatments for 5 days.

DETAILED DESCRIPTION:
Perinatal depression is underdiagnosed, undertreated, and understudied. Approximately one in five individuals will experience perinatal depression, which spans from conception to one year after birth. Untreated perinatal depression increases the risk of stillbirth, preterm birth, substance abuse, parental suicide, and developmental delay. There are limited empirical data to guide treatment of perinatal depression. Psychotherapy can be effective for mild-to-moderate depression, but it is slow acting and difficult to access. Antidepressants show inconsistent benefits and safety; moreover, patients report feeling anxious or guilty about taking them.

Transcranial magnetic stimulation (TMS) is FDA cleared treatment for major depressive disorder, adolescent depression, late life depression, and anxious depression. It has also shown promise as a safe and effective biological intervention for perinatal depression for both the mother and fetus. One of the most exciting new developments in neurostimulation is accelerated intermittent theta burst stimulation (iTBS), a TMS protocol that involves multiple daily treatments rather than once daily treatment. A specific accelerated TMS protocol called Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT) was FDA cleared in September 2022 because of its rapid and robust antidepressant effects. In an open-label study (n=21), SNT significantly reduced depression in one day and yielded 90.5% remission after five days. Importantly, there is no evidence that accelerated TMS protocols pose more risk than conventional TMS protocols that have a strong safety profile.

While SNT is a potential breakthrough treatment, it has not been tested in peripartum individuals. Accelerated iTBS may expedite depressive symptom improvement and reduce the need for pharmacotherapy for individuals struggling with perinatal depression. If tolerable and efficacious, this treatment modality may increase the viable treatment options available to peripartum women with depressive symptoms.

In this pilot trial, patients who are currently pregnant or postpartum with treatment-resistant depression (n=12) will receive a modified SNT with neuronavigation. Treatment site location will be guided by MRI when possible given the promising internal findings highlighted above. However, if neuroimaging is not chosen by the patient, unsafe for the patient for any reason, or not tolerable for the patient, we will offer treatment with scalp-based measurement (i.e., TMS targeting based on Beam F3 method). Overall, this study is critically important for informing the viability of future accelerated iTBS trials in a peripartum population and may shape the future of affective treatment options in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* All individuals must be 14-34 weeks gestational age or within one year of delivery at the time of treatment. The odds of delivery nears 10% after 36 weeks, which would limit participants from being able to complete the study and interfere with the primary study aim to understand safety and tolerability. Additionally, after 36 weeks, the standard of care is weekly obstetric check-in visits, which would be challenging for patients to complete given the time demands of the study protocol.
* Patients will not be scanned after 32 weeks gestational age due to the time needed to construct the individualized treatment target. Individuals seeking treatment beyond 32 weeks will be offered scalp-based target localization so as not to limit patient access to care.
* English proficiency sufficient for informed consent, questionnaires/tasks, and treatment
* Primary diagnosis of major depressive disorder per DSM-V criteria (MINI International Neuropsychiatric Interview/ Structured Clinical Interview for DSM-5): >20 on the Montgomery-Åsberg Depression Rating Scale (MADRS) and moderate to severe level of treatment resistance (Maudsley Staging Method)
* Stable antidepressant medication regimen, or remain medication free, for 4 weeks prior to treatment and to remain on this regimen throughout the treatment course. We request that this regimen remain stable until the 1 month post-treatment if clinically appropriate.
* Primary clinician (e.g. psychiatrist, therapist, psychologist, APRN, PA, etc.) responsible for psychiatric care before, during, and after the trial in addition to an obstetric provider responsible for obstetric care.
* Agreement to lifestyle considerations: Continue usual intake patterns of caffeine- or xanthine-containing products (e.g. coffee, tea, soft drinks, chocolate) throughout treatment

Exclusion Criteria:

* Concurrent use of rapid acting antidepressant agent (ketamine/esketamine/ECT)
* Receiving or planning to receive other TMS treatments during course of participation
* Obstetric concerns: Preeclampsia and/or current frequent, painful contractions (more than one every 10 minutes)
* History of: Neurosurgical intervention for depression, autism spectrum disorder, intellectual disability, severe cognitive impairment, significant neurological illness (e.g., dementia, Parkinson's, Huntington's, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, brain lesion), untreated or insufficiently treated endocrine disorder, and/or treatment with investigational drug or intervention during the study period
* ≥ 30% change in MADRS score between screening and baseline
* Anyone presenting with: Mania or hypomania, psychosis, active suicidal ideation with plan and some intent to act or a suicide attempt (defined by C-SSRS) within the past 3 months, neurological lesion, contraindications to either TMS or MRI (e.g., metallic implants, severe insomnia > 4 hours per night with hypnotic, etc.), and/or current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal
* Existing tinnitus (ringing in the ears) that causes functional impairment
* History of retinal detachment or other retinal pathology
* Severe borderline personality disorder
* Any other condition deemed by the PI to interfere with the study or increase risk to the participant

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability as measured by ratings of the Client Satisfaction Questionnaire (CSQ-8) | 1 month after treatment
  The CSQ-8 asks individuals about their overall experience with aTMS.Higher scores indicate a greater level of tolerability. We hypothesize that participants will report high levels of treatment satisfaction (>24) on the Client Satisfaction Questionnaire (CSQ-8).
  The primary outcome will be a composite defined as meeting 3 out of 4 metrics listed here.
Acceptability as measured by percentage of individuals who complete an entire treatment course | 1 month after treatment
  Higher percentage of individuals who completed an entire course (i.e., 50 treatments) indicates higher acceptability. We hypothesize that 9/12 participants will complete at least 75% of treatments.
  The primary outcome will be a composite defined as meeting 3 out of 4 metrics here.
Safety as measured by reports of adverse events | 1 month after treatment
  We will monitor and report the rate of serious adverse events, including maternal seizures in the sample. We hypothesize that there will be no serious adverse events.
Feasibility as measured by the number of individuals treated throughout the study | From the beginning to the end of the study
  Report of the number of individuals who received treatment throughout the entire study (i.e., approximately 2 years). We hypothesize that we will be able to enroll and treat 12 participants in two years.
  The primary outcome will be a composite defined as meeting 3 out of 4 metrics here.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | From baseline to 1 month post treatment.
  A clinician rated tool used to assess the severity of depression in adults. The MADRS consists of 10 items, each scored on a 7 point scale 0-6 with higher scores indicating more severe depressive symptoms.
Assess the effects of accelerated TMS on birth outcomes and lactation | Throughout the 5 days of treatment to 1 month post treatment
  We will monitor and report neonatal APGAR scores from infants delivered from mothers in the sample, birth weights, intradelivery maternal pain scores, birth modality (e.g. vaginal or C-section), and maternal blood loss. For individuals postpartum, we will ask participants to log their milk supply daily during treatment to determine any effects

OTHER OUTCOMES:
Beck Depression Inventory (BDI) | Before treatment, daily throughout treatment, 2 week post treatment, and 1 month post treatment
  Depression severity rating scales (0-63, higher numbers indicate higher severity)
Beck Anxiety Inventory (BAI) | Before treatment, daily throughout treatment, 2 week post treatment, and 1 month post treatment
  Anxiety severity rating scale (0-63, higher numbers indicate higher severity)
Young Mania Rating Scale (YMRS) | Before treatment, daily throughout treatment, 2 week post treatment, and 1 month post treatment
  11 item scale evaluating mania. Scored 0-60. Higher score indicates worse outcome/higher mania
Edinburgh Postnatal Depression Scale | Before treatment, 2 weeks after treatment, and 1 month after treatment.
  A scale created to help identify women who may be suffering from postpartum depression. Each question is scored 0-3, with a maximum score of 30. A score of more than 10 suggests minor or major depression may be present.
Hamilton Rating Scale for Depression | Before treatment, 2 weeks after treatment, and 1 month after treatment.
  Designed to rate the severity of depression in individuals. Scores range from 0-52, a higher score indicating more severe depression.
Maternal Ante/Postnatal Attachment Scale | Before treatment, 2 weeks after treatment, and 1 month after treatment.
  Developed to assess a new mother's emotional response to her infant. Each item is rated on a 5-point scale (typically ranging from 1 to 5). Lower scores indicate lower attachment.
PTSD Checklist with Criterion A for DSM-5 | Before treatment, 2 weeks after treatment, and 1 month after treatment.
  20 item PTSD scale, scored 0-80. Higher scores indicate worse symptoms.
Adult Temperament Questionnaire | Before treatment, 2 weeks after treatment, and 1 month after treatment.
  77-item self-report questionnaire assessing individuals temperament and personality. Scores range from 0-539, with scores in subsections of the questionnaire indicating various affects and temperaments.
Perinatal Anxiety Screening Scale | Before treatment, 2 weeks after treatment, and 1 month after treatment.
  31-item self-report instrument designed to screen for problematic anxiety in antenatal and postpartum women. Each item is rated on a 4-point Likert scale (0-4), with higher scores indicating greater anxiety.
Emotion Reactivity Scale | Before treatment, 2 weeks after treatment, and 1 month after treatment.
  21-item self-report measure designed to assess an individual's emotional reactivity. Responses are scored on a 5-point Likert scale, with higher scores indicating greater emotional reactivity.
Standford Expectations of Treatment Scale | Baseline visit
  Measures patient outcome expectancy in clinical trials, specifically focusing on positive and negative treatment expectations. Scores range from 3-21, with higher scores indicating higher belief treatment will work, lower scores indicating more skepticism/anxiety about treatment being successful.
Patient Global Impressions | Baseline, 2 weeks after treatment, 1 month after treatment
  A single question assessing a patient's perception of their health or condition. Scores range from 1-7, one being the participant believes they are not at all ill, seven being an extremely ill individual.
World Health Organization Quality of Life - Brief Version | Before treatment, 2 weeks after treatment, and 1 month after treatment.
  26-item questionnaire to assess quality of life. Uses a 5-point Likert scale, with higher scores indicating higher perceived quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided